CLINICAL TRIAL: NCT01121419
Title: The Role of IMP3 Expression in Patients With Neuroblastoma
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Wen-Ming Hsu, National Taiwan University Hospital
Other Study IDs: 201002039R
Record Dates: First submitted 2010-05-03; First posted 2010-05-12 (Estimated); Last update posted 2010-05-21 (Estimated); Status verified 2010-05

CONDITIONS: Neuroblastoma
Keywords: Neuroblastoma; IMP3; Prognosis
MeSH Terms: conditions — Neuroblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Neuroblastoma

SUMMARY:
Neuroblastoma (NB), a common cancer of early childhood originating from primitive sympathetic neural precursors, is characterized by the remarkable heterogeneity of clinical behaviors from spontaneous regression to rapid progression and death. The current therapeutic options are developed according to the Children's Oncology Group (COG) risk stratification criteria based on clinical and biological factors, including tumor stage, MYCN status, age at diagnosis, histology, and ploidy status. 1-2 The treatment strategies ranging from observation alone to intensive multimodality therapy depends on the risk stratification of three subgroups of low, intermediate, and high risk of death. Despite a number of molecular and biologic factors has been identified to predict the prognosis, MYCN amplification, which occurring in roughly 20% of primary NB, is one of the most powerful prognostic factors.3 The co-opting neurotrophin pathways including the neurotrophin receptors (TrkA, TrkB, and TrkC) and their ligands (NGF, BDNF, and neurotrophin-3, respectively), which regulate the differentiation, apoptosis, and growth of neural cells, are also important molecules related to the prognosis of NB.4 However, a proportion of patients with MYCN nonamplified NB still presents clinically aggressive progression similar to those of MYCN amplified tumors, suggesting that other unfavorable molecules exist for the inferior survival.5-6 The IGF-II RNA-binding protein 3 (IMP3), also known as L532S or K homology domain-containing protein overexpressed in cancer (KOC), is a member of RNA-binding protein family which includes IMP1, IMP2, and IMP3. The IMPs are primarily expressed during early embryogenesis and have been implicated in various post-transcriptional functions, including mRNA localization, cell growth, and cell migration during early embryogenesis.7-8 The IMP3 orthologue Vg1-RBP in Xenopus has also been described to promote migration of neural crest cells.9 Recently, the IMP3 is considered an oncofetal protein by increasing proliferation and invasion in various cancers including pancreas, kidney, and lung cancers.10-14 The expression of IMP3 is, however, low or undetectable in adjacent benign tissues.13 These lines of evidence indicate that IMP3 is capable of a potential biomarker to predict cancer progression and metastasis, and may serve as a target molecule for cancer therapy.14

oligonucleotide microarray is a powerful tool to do a genome-wide screening of candidate genes related to cancer prognosis.15 In this study, 22 primary NB tumors were subjected to oligonucleotide microarray analysis. Among the differentially expressed genes according to the patients' prognosis, IMP3 showed an especially high expression level in NB tumors carrying unfavorable prognosis. Further evaluation of IMP3 expression in a large sample size demonstrated that IMP3 expression could predict an unfavorable prognosis of NB patients independent of other biomarkers. Targeting of IMP3 expression in a NB cell line did suppress cell invasion ability, suggesting that IMP3 could not only be a prognostic factor, but also be a potential therapeutic target of NB.

ELIGIBILITY:
Inclusion Criteria:

* Neuroblastoma patients with complete follow-up and sufficient samples for study.

Exclusion Criteria:

* Neuroblastoma patients without complete follow-up
* Neuroblastoma patients without sufficient samples for study.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: From January 1990 to December 2009, 90 pediatric patients of NB treated at the National Taiwan University Hospital, Taiwan
Sampling Method: Non-Probability Sample
Dates: Start 2008-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Ming Hsu, M.D, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Wen-Ming Hsu, Taipei, Taiwan